CLINICAL TRIAL: NCT03927534
Title: Efficacy of a Mindful Eating Program to Reduce Emotional Eating in Patients Suffering From Overweight or Obesity in Primary Care Settings: a Cluster Randomized Controlled Clinical Trial Protocol
Brief Title: Efficacy of a Mindful-eating Program to Reduce Emotional Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Dharamsala Institute of Mindfulness and Psychotherapy of Zaragoza (Unknown)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/2019
Record Dates: First submitted 2019-04-19; First posted 2019-04-25 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Overweight; Mindful Eating; Primary Care; Randomized controlled trial (RCT)
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Mindful Eating program is apply face to face 7 sessions of 120 minutes/session. ME is apply in groups of 10-12 people in traditional format. Written material and sound recordings will be offered as support elements. The estimated duration of the face to face program is two months.
  Interventions: Behavioral: Mindful Eating
- Control (No Intervention): Treatment As Usual (TAU) in Primary Care (PC) is any kind of treatment administered by the GP to the patient with overweight and obesity. According to nutritional status, overweight or obesity, as well as the presence of co-morbidity, different actions can comprise the treatment offered at a PC level. For individuals presenting with overweight (BMI 25-29.9 kg/m2) but with no co-morbidities, PC teams organise care plans to enable them to achieve a normal BMI range (BMI 18.5-24.9 kg/m2). In case of suicide risk, severe social dysfunction or worsening of symptoms, it is recommended that patients are referred to mental health facilities.

INTERVENTIONS:
Behavioral: Mindful Eating — The ME group will be composed by 7 weekly group sessions with a minimum duration of two hours, mixing theoretical contents with practices. Sessions will always be the same day of the week, except for bank holidays or eventualities, and will be conducted by a psychologist specially trained and certified in ME with experience in leading mindfulness groups. Group sizes will range between 10 and 12 participants. At the end of each session, participants will receive theoretical contents and homework activities to be practiced along the week.
  Arms: Experimental

SUMMARY:
Mindfulness-Based Interventions have been applied in different fields to improve physical and psychological health. However, little is known about its applicability and effectiveness in Spanish adults with overweight and obesity. The aim of the present study protocol is to evaluate the feasibility and efficacy of an adapted MBI programme to reduce emotional eating in adults with overweight and obesity in primary care (PC) settings.

DETAILED DESCRIPTION:
This study is a multi-centre, two-armed randomized controlled trial (RCT), with pre-treatment, post-treatment and 1-year follow-up measures, and a 1:1 allocation rate between groups. Patients from four mental health units in Zaragoza (Spain) will be randomly assigned to two different parallel conditions, with one psychological intervention group ('ME + TAU') and usual treatment ('TAU alone') managed by their general practitioner (GP), to test the superiority of 'ME + TAU' provision compared with 'TAU alone' provision. For ethical reasons, those patients allocated to 'TAU alone' will be offered the ME programme after finishing the trial at 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45-75 years
* Have overweight or obesity condition based in BMI (Body Mass Index). Individuals with BMI of 25 or more.
* Have two of these three risk: sedentary lifestyle, poor diet and binge episodes.
* Ability to understand oral and written Spanish.
* Willingness to participate in the study and signing informed consent.

Exclusion Criteria:

* Any diagnosis of a disease that may affect the central nervous system (brain condition, traumatic brain injury, dementia, etc).
* Other psychiatric diagnoses or acute psychiatric illness (substance dependence or abuse, history of schizophrenia or other psychotic disorders, etc.), except for anxiety disorder or personality disorders.
* Presence of delusional ideas or hallucinations whether consistent or not with mood.
* Suicide risk.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
The Dutch Eating Behavior Questionnaire | Baseline in experimental and control groups.
  It was designed to measure eating styles that may attenuate or contribute to the development of overweight. It comprises three scales that measure emotional, external and restrained eating. The Spanish version of the DEBQ has 33 items, 13 of them referred to the emotional eating scale (e.g., "Desire to eat when irritated"), and 10 items referring to the external (e.g., "Eating when you feel lonely") and restrictive (e.g., "Difficult to resist delicious food") scales, respectively. The items can be rated on a five-point likert scale with 1 indicating "never" and 5 indicating "very often".
The Dutch Eating Behavior Questionnaire | Post-treatment 8 weeks from baseline in experimental and control groups
  It was designed to measure eating styles that may attenuate or contribute to the development of overweight. It comprises three scales that measure emotional, external and restrained eating. The Spanish version of the DEBQ has 33 items, 13 of them referred to the emotional eating scale (e.g., "Desire to eat when irritated"), and 10 items referring to the external (e.g., "Eating when you feel lonely") and restrictive (e.g., "Difficult to resist delicious food") scales, respectively. The items can be rated on a five-point likert scale with 1 indicating "never" and 5 indicating "very often".
The Dutch Eating Behavior Questionnaire | twelve-months follow-up in experimental and control groups
  It was designed to measure eating styles that may attenuate or contribute to the development of overweight. It comprises three scales that measure emotional, external and restrained eating. The Spanish version of the DEBQ has 33 items, 13 of them referred to the emotional eating scale (e.g., "Desire to eat when irritated"), and 10 items referring to the external (e.g., "Eating when you feel lonely") and restrictive (e.g., "Difficult to resist delicious food") scales, respectively. The items can be rated on a five-point likert scale with 1 indicating "never" and 5 indicating "very often".

SECONDARY OUTCOMES:
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline in experimental and control groups
Five Facet Mindfulness Questionnaire | Baseline in experimental and control groups
  The FFMQ-short form is a 24-item questionnaire that measures five aspects of mindfulness and there is a Spanish version based on it with appropriate psychometrics. The five facets the FFMQ measures are: observing (α = 81), describing (α = .87), acting with awareness (5 items, α = .83), non-judging to (5 items, α = .83) and non-reacting of (5 items, α = .75) inner experience. The participants indicate on a 5-point Likert scale the degree in which each item is generally true for them, ranging from 1 ("never or very rarely true") to 5 ("very often or always true").
Five Facet Mindfulness Questionnaire | Post-treatment 8 weeks from baseline in experimental and control groups
  The FFMQ-short form is a 24-item questionnaire that measures five aspects of mindfulness and there is a Spanish version based on it with appropriate psychometrics. The five facets the FFMQ measures are: observing (α = 81), describing (α = .87), acting with awareness (5 items, α = .83), non-judging to (5 items, α = .83) and non-reacting of (5 items, α = .75) inner experience. The participants indicate on a 5-point Likert scale the degree in which each item is generally true for them, ranging from 1 ("never or very rarely true") to 5 ("very often or always true").
Five Facet Mindfulness Questionnaire | twelve-months follow-up in experimental and control groups
  The FFMQ-short form is a 24-item questionnaire that measures five aspects of mindfulness and there is a Spanish version based on it with appropriate psychometrics. The five facets the FFMQ measures are: observing (α = 81), describing (α = .87), acting with awareness (5 items, α = .83), non-judging to (5 items, α = .83) and non-reacting of (5 items, α = .75) inner experience. The participants indicate on a 5-point Likert scale the degree in which each item is generally true for them, ranging from 1 ("never or very rarely true") to 5 ("very often or always true").
Self-Compassion Scale | Baseline in experimental and control groups
  It is the most used self-report instrument to measure self-compassion and it is divided into six subscales: Self-Kindness; Self-Judgment; Common Humanity; Isolation; Mindfulness; and Over-Identification. The items can be rated on a five-point Likert-type scale with 1 indicating "almost never" and 5 indicating "almost always". After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion
Self-Compassion Scale | Post-treatment 8 weeks from baseline in experimental and control groups
  It is the most used self-report instrument to measure self-compassion and it is divided into six subscales: Self-Kindness; Self-Judgment; Common Humanity; Isolation; Mindfulness; and Over-Identification. The items can be rated on a five-point Likert-type scale with 1 indicating "almost never" and 5 indicating "almost always". After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion
Self-Compassion Scale | twelve-months follow-up in experimental and control groups
  It is the most used self-report instrument to measure self-compassion and it is divided into six subscales: Self-Kindness; Self-Judgment; Common Humanity; Isolation; Mindfulness; and Over-Identification. The items can be rated on a five-point Likert-type scale with 1 indicating "almost never" and 5 indicating "almost always". After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion
Mindful Eating Scale | Baseline in experimental and control groups
  The MES scale has 28 items, including six factors: acceptance (α = .89), awareness (α = .82), non-reactivity (α = .77), act with awareness (α = .81), routine (α = .75) and unstructured eating (α = .60). Items can be rated on a 4-point Likert-type scale, with 1 indicating "never" and 4 indicating "very often".
Mindful Eating Scale | Post-treatment 8 weeks from baseline in experimental and control groups
  The MES scale has 28 items, including six factors: acceptance (α = .89), awareness (α = .82), non-reactivity (α = .77), act with awareness (α = .81), routine (α = .75) and unstructured eating (α = .60). Items can be rated on a 4-point Likert-type scale, with 1 indicating "never" and 4 indicating "very often".
Mindful Eating Scale | twelve-months follow-up in experimental and control groups
  The MES scale has 28 items, including six factors: acceptance (α = .89), awareness (α = .82), non-reactivity (α = .77), act with awareness (α = .81), routine (α = .75) and unstructured eating (α = .60). Items can be rated on a 4-point Likert-type scale, with 1 indicating "never" and 4 indicating "very often".
Bulimic Investigatory Test | Baseline in experimental and control groups
  The BITE is very used to measure the presence and severity of bulimic symptoms in nonclinical samples. Normative values for BITE total and sub-scale scores in clinical and non-clinical samples are reported. The scale includes in the Symptoms subscale (30 yes-no items; range =0-30) and Severity subscale (6 dimensional items addressing specific bulimic behaviors; range=0-39). In addition to these standars scores, another measure was derived from the BITE-the reported frequency of bingeing
Bulimic Investigatory Test | Post-treatment 8 weeks from baseline in experimental and control groups
  The BITE is very used to measure the presence and severity of bulimic symptoms in nonclinical samples. Normative values for BITE total and sub-scale scores in clinical and non-clinical samples are reported. The scale includes in the Symptoms subscale (30 yes-no items; range =0-30) and Severity subscale (6 dimensional items addressing specific bulimic behaviors; range=0-39). In addition to these standars scores, another measure was derived from the BITE-the reported frequency of bingeing
Bulimic Investigatory Test | twelve-months follow-up in experimental and control groups
  The BITE is very used to measure the presence and severity of bulimic symptoms in nonclinical samples. Normative values for BITE total and sub-scale scores in clinical and non-clinical samples are reported. The scale includes in the Symptoms subscale (30 yes-no items; range =0-30) and Severity subscale (6 dimensional items addressing specific bulimic behaviors; range=0-39). In addition to these standars scores, another measure was derived from the BITE-the reported frequency of bingeing
Eating Attitude test (EAT-26) | Baseline in experimental and control groups
  The EAT-26 had three subscales Dieting, Bulimia and Food Preocupation, and Oral Control. It is and abbreviated version of the original EAT-40, having an excellent correlation. In the EAT-26 each item is answered on a 6-point Lickert scale and if the scoring is 20 or higher the patient should look for professional advice. The Eat-26 had an elevated reliability
Eating Attitude test (EAT-26) | Post-treatment 8 weeks from baseline in experimental and control groups
  The EAT-26 had three subscales Dieting, Bulimia and Food Preocupation, and Oral Control. It is and abbreviated version of the original EAT-40, having an excellent correlation. In the EAT-26 each item is answered on a 6-point Lickert scale and if the scoring is 20 or higher the patient should look for professional advice. The Eat-26 had an elevated reliability
Eating Attitude test (EAT-26) | twelve-months follow-up in experimental and control groups
  The EAT-26 had three subscales Dieting, Bulimia and Food Preocupation, and Oral Control. It is and abbreviated version of the original EAT-40, having an excellent correlation. In the EAT-26 each item is answered on a 6-point Lickert scale and if the scoring is 20 or higher the patient should look for professional advice. The Eat-26 had an elevated reliability
Weight | Baseline in experimental and control groups
  Weight measurement will be quantified in kilograms using a digital scale
Weight | twelve-months follow-up in experimental and control groups
  Weight measurement will be quantified in kilograms using a digital scale
Abdominal perimeter | Baseline in experimental and control groupsw-up in experimental and control groups
  Abdominal perimeter measurement will be quantified in centimetres using a measuring tape
Abdominal perimeter | twelve-months follow-up in experimental and control groups
  Abdominal perimeter measurement will be quantified in centimetres using a measuring tape
Height | Baseline in experimental and control groups
  Height measurement will be quantified in centimetres using a measuring tape
Height | twelve-months follow-up in experimental and control groups
  Height measurement will be quantified in centimetres using a measuring tape
Cholesterol total | Baseline in experimental and control groups
  Cholesterol total measurement will be quantified mg/dL using a blood test
Cholesterol total | twelve-months follow-up in experimental and control groups
  Cholesterol total measurement will be quantified mg/dL using a blood test
LDL | Baseline in experimental and control groups
  LDL measurement will be quantified mg/dL using a blood test
LDL | twelve-months follow-up in experimental and control groups
  LDL measurement will be quantified mg/dL using a blood test
HDL | Baseline in experimental and control groups
  HDL measurement will be quantified mg/dL using a blood test
HDL | twelve-months follow-up in experimental and control groups
  HDL measurement will be quantified mg/dL using a blood test
Glucose | Baseline in experimental and control groups
  Glucose measurement will be quantified mg/dL using a blood test
Glucose | twelve-months follow-up in experimental and control groups
  Glucose measurement will be quantified mg/dL using a blood test
Alanine aminotransferase | Baseline in experimental and control groups
  Alanine aminotransferase measurement will be quantified U/L using a blood test
Alanine aminotransferase | twelve-months follow-up in experimental and control groups
  Alanine aminotransferase measurement will be quantified U/L using a blood test
Glycated haemoglobin | Baseline in experimental and control groups
  Glycated haemoglobin measurement will be quantified in percentage (%) using a blood test
Glycated haemoglobin | twelve-months follow-up in experimental and control groups
  Glycated haemoglobin measurement will be quantified in percentage (%) using a blood test
General Anxiety Disorder | Baseline in experimental and control groups
  It is one of the most frequently used diagnostic self-report scales for screening, diagnosis and anxiety disorder severity assessment, defined as an excessive anxiety and worry (apprehensive expectation) related to a number of events or activities, associated to experiencing difficulties to control that worry. Items are rated on a 4-point Likert-type scale (between 0 = "not at all" and 3 = "nearly every day"). The GAD-7 inquires about events happening over the last two weeks, in order to know how often the patient has been bothered by them
General Anxiety Disorder | twelve-months follow-up in experimental and control groups
  It is one of the most frequently used diagnostic self-report scales for screening, diagnosis and anxiety disorder severity assessment, defined as an excessive anxiety and worry (apprehensive expectation) related to a number of events or activities, associated to experiencing difficulties to control that worry. Items are rated on a 4-point Likert-type scale (between 0 = "not at all" and 3 = "nearly every day"). The GAD-7 inquires about events happening over the last two weeks, in order to know how often the patient has been bothered by them
Patient Health Questionnaire | Baseline in experimental and control groups
  This scale is one of the most widely used questionnaires that assess the intensity of depression in pharmacological and psychological studies, it is useful to monitor changes experienced by patients over time. Through items like "Little interest or pleasure in doing things" and using a Liker-type scale from 0 ("not at all") to 3 ("nearly every day"), the PHQ-9 reflects the experience of participants during the last two weeks.
Patient Health Questionnaire | twelve-months follow-up in experimental and control groups
  This scale is one of the most widely used questionnaires that assess the intensity of depression in pharmacological and psychological studies, it is useful to monitor changes experienced by patients over time. Through items like "Little interest or pleasure in doing things" and using a Liker-type scale from 0 ("not at all") to 3 ("nearly every day"), the PHQ-9 reflects the experience of participants during the last two weeks.
The diastolic blood pressure (DBP) and the systolic blood pressure (SBP) | Baseline in experimental and control groups
  In order to evaluate the vital signs we will use a vascular screening system, in the version VaSera VS-1500.
The diastolic blood pressure (DBP) and the systolic blood pressure (SBP) | twelve-months follow-up in experimental and control groups
  In order to evaluate the vital signs we will use a vascular screening system, in the version VaSera VS-1500.

CONTACTS AND LOCATIONS:
Overall Officials: Javier García-Campayo, PhD, Principal Investigator — Miguel Servet Hospital and University of Zaragoza
Locations (1):
- Department of Psychiatry. Miguel Servet University Hospital, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Once available, the results of the trial will be presented at national and international conferences and in peer-reviewed journal publications. Due to the clinical nature of the study and considering ethical concerns, the data (anonymised and completely de-identified) generated by this trial will be made available upon request to researchers a) who provide a methodologically sound proposal and b) whose proposed use of the data has been approved by an independent ethical review committee. Data will become available following each publication with no end date for replicating the results of the trial or for any analytical purpose that is related to achieve aims in the original proposal. The database will be encrypted and password protected (passwords will be provided by the corresponding author to researchers that meet the referred criteria).
Time Frame: Data will become available following each publication with no end date for replicating the results of the trial or for any analytical purpose
Access Criteria: Due to the clinical nature of the study and considering ethical concerns, the data (anonymised and completely de-identified) generated by this trial will be made available upon request to researchers a) who provide a methodologically sound proposal and b) whose proposed use of the data has been approved by an independent ethical review committee
URL: http://doi.org/10.3886/E111741V1

REFERENCES:
- [Background] Rossner S. Obesity: the disease of the twenty-first century. Int J Obes Relat Metab Disord. 2002 Dec;26 Suppl 4:S2-4. doi: 10.1038/sj.ijo.0802209. PMID 12457290
- [Background] Mann T, Tomiyama AJ, Westling E, Lew AM, Samuels B, Chatman J. Medicare's search for effective obesity treatments: diets are not the answer. Am Psychol. 2007 Apr;62(3):220-33. doi: 10.1037/0003-066X.62.3.220. PMID 17469900
- [Background] Holzel BK, Lazar SW, Gard T, Schuman-Olivier Z, Vago DR, Ott U. How Does Mindfulness Meditation Work? Proposing Mechanisms of Action From a Conceptual and Neural Perspective. Perspect Psychol Sci. 2011 Nov;6(6):537-59. doi: 10.1177/1745691611419671. PMID 26168376
- [Background] Kristeller JL, Hallett CB. An Exploratory Study of a Meditation-based Intervention for Binge Eating Disorder. J Health Psychol. 1999 May;4(3):357-63. doi: 10.1177/135910539900400305. PMID 22021603
- [Background] Medina WL, Wilson D, de Salvo V, Vannucchi B, de Souza EL, Lucena L, Sarto HM, Modrego-Alarcon M, Garcia-Campayo J, Demarzo M. Effects of Mindfulness on Diabetes Mellitus: Rationale and Overview. Curr Diabetes Rev. 2017;13(2):141-147. doi: 10.2174/1573399812666160607074817. PMID 27280721
- [Background] Rosenzweig S, Reibel DK, Greeson JM, Edman JS, Jasser SA, McMearty KD, Goldstein BJ. Mindfulness-based stress reduction is associated with improved glycemic control in type 2 diabetes mellitus: a pilot study. Altern Ther Health Med. 2007 Sep-Oct;13(5):36-8. PMID 17900040
- [Background] Miller CK, Kristeller JL, Headings A, Nagaraja H, Miser WF. Comparative effectiveness of a mindful eating intervention to a diabetes self-management intervention among adults with type 2 diabetes: a pilot study. J Acad Nutr Diet. 2012 Nov;112(11):1835-42. doi: 10.1016/j.jand.2012.07.036. PMID 23102183
- [Background] Fanning J, Osborn CY, Lagotte AE, Mayberry LS. Relationships between dispositional mindfulness, health behaviors, and hemoglobin A1c among adults with type 2 diabetes. J Behav Med. 2018 Dec;41(6):798-805. doi: 10.1007/s10865-018-9938-3. Epub 2018 May 25. PMID 29802533
- [Background] Mantzios M, Wilson JC. Mindfulness, Eating Behaviours, and Obesity: A Review and Reflection on Current Findings. Curr Obes Rep. 2015 Mar;4(1):141-6. doi: 10.1007/s13679-014-0131-x. PMID 26627097
- [Background] Godsey J. The role of mindfulness based interventions in the treatment of obesity and eating disorders: an integrative review. Complement Ther Med. 2013 Aug;21(4):430-9. doi: 10.1016/j.ctim.2013.06.003. Epub 2013 Jul 9. PMID 23876574
- [Background] Mason AE, Epel ES, Kristeller J, Moran PJ, Dallman M, Lustig RH, Acree M, Bacchetti P, Laraia BA, Hecht FM, Daubenmier J. Effects of a mindfulness-based intervention on mindful eating, sweets consumption, and fasting glucose levels in obese adults: data from the SHINE randomized controlled trial. J Behav Med. 2016 Apr;39(2):201-13. doi: 10.1007/s10865-015-9692-8. Epub 2015 Nov 12. PMID 26563148
- [Derived] Morillo Sarto H, Barcelo-Soler A, Herrera-Mercadal P, Pantilie B, Navarro-Gil M, Garcia-Campayo J, Montero-Marin J. Efficacy of a mindful-eating programme to reduce emotional eating in patients suffering from overweight or obesity in primary care settings: a cluster-randomised trial protocol. BMJ Open. 2019 Nov 21;9(11):e031327. doi: 10.1136/bmjopen-2019-031327. PMID 31753880